CLINICAL TRIAL: NCT03711682
Title: Hypoglycemic Effect of Cinnamomum Verum in Type 2 Diabetic Patients in the Municipality of Comasagua
Brief Title: Reducing Plasma Glucose Effect of Cinnamon in Type 2 Diabetic Patients in the Municipality of Comasagua
Acronym: GCIG
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Dr. José Matías Delgado (Other)
Collaborators: Hospital Nacional Rosales (Other); Unidad Comunitaria de Salud Familiar Intermedia de Comasagua (UCSFI-Comasagua) (Unknown); Asociación Salvadoreña de Diabetes (ASADI) (Unknown)
Responsible Party: Principal Investigator, Miguel Antonio Padilla Pimentel, MD, Doctor of Medicine, Universidad Dr. José Matías Delgado
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-2017
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Glucose; Cinnamomum verum; Cinnamomum zeylanicum; Cinnamon; HbA1c; Blood Pressure; Glycated Hemoglobin; Diastolic Pressure; Systolic Pressure; Body Mass Index; BMI; Metformin; Waist Circumference
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon (Intervented) (Experimental)
  Interventions: Dietary Supplement: Cinnamon
- Wheat Flour (Placebo) (Placebo Comparator)
  Interventions: Dietary Supplement: Wheat Flour

INTERVENTIONS:
Dietary Supplement: Cinnamon — Participants in this group will receive cinnamon capsules for 12 weeks period. With a 2 g dose in capsules with 500 mg of cinnamon powder (Cinnamomum verum), 1 g in during the breakfast (2 capsules) and the other 1 g (2 capsules) during the dinner.
  Other Names: Intervened; Group A
  Arms: Cinnamon (Intervented)
Dietary Supplement: Wheat Flour — Participants in this group will receive placebo capsules for 12 weeks period. With a 2 g dose in capsules with 500 mg of wheat flour(fortified with iron, niacin, thiamin, riboflavin and folic acid), 1 g in during the breakfast (2 capsules) and the other 1 g (2 capsules) during the dinner.
  Other Names: Placebo; Group B
  Arms: Wheat Flour (Placebo)

SUMMARY:
The aim of the study is evaluate the effect of cinnamon powder (Cinnamomum verum) on the glycaemia and HbA1c (Glycohemoglobin) of type 2 diabetic Salvadoran patients, whose hypoglycemic treatment is only Metformin. To carry out this objective, subjects who agree to be part of the study will subjected to measurements of their body weight, height, body mass index, waist circumference, systolic pressure, diastolic pressure, capillary glucose (with glucose meter) every 2 weeks, and their glycohemoglobin (HbA1c) at the beginning and at the end of the study.

DETAILED DESCRIPTION:
The study will be conducted for 12 weeks (3 months) with 30 participants diagnosed with type 2 diabetes mellitus, whose only treatment for diabetes is metformin.

Both, intervention with Cinnamon (Cinnamomum verum) and wheat flour (placebo) will be encapsulated in titanium white capsules with 500 mg of powder, that will take place in agro-industry laboratories, and will be packed in glass bottles with a content of 56 capsules and a bag of silica gel.

The data of the probable participants will verified with their medical records in the Intermediate Communitarian Unit of Family Health of Comasagua municipality (UCSFI-Comasagua). Then those who meet the criteria will contacted to be enrolled in the study, if they agreed, an informed consent will signed or stamped if the participant cannot read and write.

The randomization will be make using a list of the participants and them using the Graphpad QuickCalcs option of "Randomly assign participants to groups", assigning the participants to a group A (intervention) or B (placebo).

Participants in both groups will continue to receive the treatment they would normally receive from their respective primary care providers during the duration of the study.

The participants, who accepted and signed the informed consent, will provided with a moth calendar with the schedule of the measures. The measured variables are body weight, height, body mass index, waist circumference, systolic pressure, diastolic pressure, capillary glucose (with glucose meter) and HbA1c. The measurements will take place every 2 weeks (week 0, 2, 4, 6, 8, 10 and 12) with the exception of HbA1c which will be measured at the beginning and at the end of the study (week 0 and 12).

The obtained data will be write in the paper medical records of each participant and then exported to a database in Microsoft Excel, after that data will processed in statistical software. In case of adverse effects, this will recorded into a formulary dedicated to it, this provided to the UCSFI-Comasagua physicians with the contact data of the researchers. In addition, to perform this study the researchers make an agreement with the UCSFI-Comasagua and with the endocrinology service of the Rosales National Hospital along with the Salvadoran Association of Diabetes (ASADI) to provide health care and support to those participants who presented adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes mellitus.
* Treated only with Metformin as unique treatment for diabetes.

Exclusion Criteria:

* Hypersensitivity or allergy reported to Cinnamomum spp. or Peruvian balm.
* Ulcer of gastrointestinal location.
* Chronic treatment with analgesics, antibiotics, estrogens, antineoplastics, antihypertensives of the beta-blocker type, anti-inflammatory, medications whose route of action is Gamma-Aminobutyric Acid and / or anticoagulants.
* Under treatment with steroid and / or aspirin.
* Subject that use alternative medicine treatments.
* Women of childbearing age who do not use any contraceptive method.
* Subjects subjected to surgical procedures in the 6 weeks prior to the beginning of the study.
* Subjects who presented fasting glycemia levels greater than 400 mg/dL in the previous control.
* Allergies to wheat and/or diagnosed with celiac disease.
* Adverse Drug Reaction during the study.
* Subjects whose treatment schedule changed during the study intervention.
* Subjects that does not accept to be part of the study, decides to leave the study or does not have adherence to the treatment provided.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Week 0 and 12

SECONDARY OUTCOMES:
Change in Capillary Glucose | Week 0, 2, 4, 6, 8, 10, 12
Change in Body Mass Index (BMI) | Week 0, 2, 4, 6, 8, 10, 12
Change in Waist Circumference | Week 0, 2, 4, 6, 8, 10, 12
Change in Diastolic pressure | Week 0, 2, 4, 6, 8, 10, 12
Change in Systolic Pressure | Week 0, 2, 4, 6, 8, 10, 12

OTHER OUTCOMES:
Change in Theoretical HbA1c | Week 0, 4, 8, 12
  Theoretical HbA1c, calculated using the mean of the capillary glucose of each month (every 4 weeks), and the formula A1c% = (AG mg/dL + 46.7) / 28.7

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Padilla, M.D., Principal Investigator — Universidad Dr. José Matías Delgado; Ana E Centeno, M.D., Principal Investigator — Universidad Dr. José Matías Delgado; Melissa V Abarca, M.D., Principal Investigator — Universidad Dr. José Matías Delgado; Roberto W Cerritos, M.D., Study Chair — Universidad de El Salvador, Hospital Nacional Rosales; William A Hoyos, M.D., Principal Investigator — Universidad Dr. José Matías Delgado; Karla M Navarrete, M.D., MPh., Principal Investigator — Secretaría Antidrogas de la Ciudad de San Salvador
Locations (1):
- Unidad Comunitaria de Salud Familiar Intermedia de Comasagua (UCSFI-Comasagua), Comasagua, La Libertad Department, El Salvador

IPD SHARING:
Plan to Share IPD: No
There's not Individual Patient Data sharing plan because at the moment the participants signed the informed consent it stipulate their individual data will not be shared.

REFERENCES:
- [Background] Medagama AB. The glycaemic outcomes of Cinnamon, a review of the experimental evidence and clinical trials. Nutr J. 2015 Oct 16;14:108. doi: 10.1186/s12937-015-0098-9. PMID 26475130
- [Background] Cramer JA. A systematic review of adherence with medications for diabetes. Diabetes Care. 2004 May;27(5):1218-24. doi: 10.2337/diacare.27.5.1218. PMID 15111553
- [Background] American Diabetes Association; Bantle JP, Wylie-Rosett J, Albright AL, Apovian CM, Clark NG, Franz MJ, Hoogwerf BJ, Lichtenstein AH, Mayer-Davis E, Mooradian AD, Wheeler ML. Nutrition recommendations and interventions for diabetes: a position statement of the American Diabetes Association. Diabetes Care. 2008 Jan;31 Suppl 1:S61-78. doi: 10.2337/dc08-S061. No abstract available. PMID 18165339
- [Background] Yeh GY, Eisenberg DM, Kaptchuk TJ, Phillips RS. Systematic review of herbs and dietary supplements for glycemic control in diabetes. Diabetes Care. 2003 Apr;26(4):1277-94. doi: 10.2337/diacare.26.4.1277. PMID 12663610
- [Background] American Diabetes Association. (2) Classification and diagnosis of diabetes. Diabetes Care. 2015 Jan;38 Suppl:S8-S16. doi: 10.2337/dc15-S005. No abstract available. PMID 25537714
- [Background] Ros Perez M, Medina-Gomez G. [Obesity, adipogenesis and insulin resistance]. Endocrinol Nutr. 2011 Aug-Sep;58(7):360-9. doi: 10.1016/j.endonu.2011.05.008. Epub 2011 Jul 22. Spanish. PMID 21778123
- [Background] Canivell S, Gomis R. Diagnosis and classification of autoimmune diabetes mellitus. Autoimmun Rev. 2014 Apr-May;13(4-5):403-7. doi: 10.1016/j.autrev.2014.01.020. Epub 2014 Jan 11. PMID 24424179
- [Background] Unoki H, Takahashi A, Kawaguchi T, Hara K, Horikoshi M, Andersen G, Ng DP, Holmkvist J, Borch-Johnsen K, Jorgensen T, Sandbaek A, Lauritzen T, Hansen T, Nurbaya S, Tsunoda T, Kubo M, Babazono T, Hirose H, Hayashi M, Iwamoto Y, Kashiwagi A, Kaku K, Kawamori R, Tai ES, Pedersen O, Kamatani N, Kadowaki T, Kikkawa R, Nakamura Y, Maeda S. SNPs in KCNQ1 are associated with susceptibility to type 2 diabetes in East Asian and European populations. Nat Genet. 2008 Sep;40(9):1098-102. doi: 10.1038/ng.208. PMID 18711366
- [Background] Chen L, Magliano DJ, Zimmet PZ. The worldwide epidemiology of type 2 diabetes mellitus--present and future perspectives. Nat Rev Endocrinol. 2011 Nov 8;8(4):228-36. doi: 10.1038/nrendo.2011.183. PMID 22064493
- [Background] Ye J. Mechanisms of insulin resistance in obesity. Front Med. 2013 Mar;7(1):14-24. doi: 10.1007/s11684-013-0262-6. Epub 2013 Mar 9. PMID 23471659
- [Background] Sacks DB. Measurement of hemoglobin A(1c): a new twist on the path to harmony. Diabetes Care. 2012 Dec;35(12):2674-80. doi: 10.2337/dc12-1348. No abstract available. PMID 23173136
- [Background] Sacks DB. Correlation between hemoglobin A1c (HbA1c) and average blood glucose: can HbA1c be reported as estimated blood glucose concentration? J Diabetes Sci Technol. 2007 Nov;1(6):801-3. doi: 10.1177/193229680700100602. No abstract available. PMID 19885151
- [Background] Unnikrishnan R, Anjana RM, Mohan V. Drugs affecting HbA1c levels. Indian J Endocrinol Metab. 2012 Jul;16(4):528-31. doi: 10.4103/2230-8210.98004. PMID 22837911
- [Background] Tancredi M, Rosengren A, Svensson AM, Kosiborod M, Pivodic A, Gudbjornsdottir S, Wedel H, Clements M, Dahlqvist S, Lind M. Excess Mortality among Persons with Type 2 Diabetes. N Engl J Med. 2015 Oct 29;373(18):1720-32. doi: 10.1056/NEJMoa1504347. PMID 26510021
- [Background] Guthrie RA, Guthrie DW. Pathophysiology of diabetes mellitus. Crit Care Nurs Q. 2004 Apr-Jun;27(2):113-25. doi: 10.1097/00002727-200404000-00003. PMID 15137354
- [Background] Johnson AM, Olefsky JM. The origins and drivers of insulin resistance. Cell. 2013 Feb 14;152(4):673-84. doi: 10.1016/j.cell.2013.01.041. PMID 23415219
- [Background] Saltiel AR, Kahn CR. Insulin signalling and the regulation of glucose and lipid metabolism. Nature. 2001 Dec 13;414(6865):799-806. doi: 10.1038/414799a. PMID 11742412
- [Background] Pessin JE, Saltiel AR. Signaling pathways in insulin action: molecular targets of insulin resistance. J Clin Invest. 2000 Jul;106(2):165-9. doi: 10.1172/JCI10582. No abstract available. PMID 10903329
- [Background] Nathan DM, Kuenen J, Borg R, Zheng H, Schoenfeld D, Heine RJ; A1c-Derived Average Glucose Study Group. Translating the A1C assay into estimated average glucose values. Diabetes Care. 2008 Aug;31(8):1473-8. doi: 10.2337/dc08-0545. Epub 2008 Jun 7. PMID 18540046
- [Background] van 't Riet E, Alssema M, Rijkelijkhuizen JM, Kostense PJ, Nijpels G, Dekker JM. Relationship between A1C and glucose levels in the general Dutch population: the new Hoorn study. Diabetes Care. 2010 Jan;33(1):61-6. doi: 10.2337/dc09-0677. Epub 2009 Oct 6. PMID 19808928
- [Background] Bonora E, Calcaterra F, Lombardi S, Bonfante N, Formentini G, Bonadonna RC, Muggeo M. Plasma glucose levels throughout the day and HbA(1c) interrelationships in type 2 diabetes: implications for treatment and monitoring of metabolic control. Diabetes Care. 2001 Dec;24(12):2023-9. doi: 10.2337/diacare.24.12.2023. PMID 11723077
- [Background] Rohlfing CL, Wiedmeyer HM, Little RR, England JD, Tennill A, Goldstein DE. Defining the relationship between plasma glucose and HbA(1c): analysis of glucose profiles and HbA(1c) in the Diabetes Control and Complications Trial. Diabetes Care. 2002 Feb;25(2):275-8. doi: 10.2337/diacare.25.2.275. PMID 11815495
- [Background] B. K. M. Goud, B. Nayal, O. S. Devi, T. G. Sathisha, S. Shivashanker and R. N. Devaki. Relation of calculated HbA1C with fasting plasma glucose and duration of diabetes. International Journal of Applied Biology and Pharmaceutical Technology. 2011;2(2):58-61.
- [Background] Dugoua JJ, Seely D, Perri D, Cooley K, Forelli T, Mills E, Koren G. From type 2 diabetes to antioxidant activity: a systematic review of the safety and efficacy of common and cassia cinnamon bark. Can J Physiol Pharmacol. 2007 Sep;85(9):837-47. doi: 10.1139/Y07-080. PMID 18066129
- [Background] Di Lorenzo C, Ceschi A, Kupferschmidt H, Lude S, De Souza Nascimento E, Dos Santos A, Colombo F, Frigerio G, Norby K, Plumb J, Finglas P, Restani P. Adverse effects of plant food supplements and botanical preparations: a systematic review with critical evaluation of causality. Br J Clin Pharmacol. 2015 Apr;79(4):578-92. doi: 10.1111/bcp.12519. PMID 25251944
- [Background] Ulbricht C, Seamon E, Windsor RC, Armbruester N, Bryan JK, Costa D, Giese N, Gruenwald J, Iovin R, Isaac R, Serrano JM, Tanguay-Colucci S, Weissner W, Yoon H, Zhang J. An evidence-based systematic review of cinnamon (Cinnamomum spp.) by the Natural Standard Research Collaboration. J Diet Suppl. 2011 Dec;8(4):378-454. doi: 10.3109/19390211.2011.627783. PMID 22432776
- [Background] Sahib AS. Anti-diabetic and antioxidant effect of cinnamon in poorly controlled type-2 diabetic Iraqi patients: A randomized, placebo-controlled clinical trial. J Intercult Ethnopharmacol. 2016 Feb 21;5(2):108-13. doi: 10.5455/jice.20160217044511. eCollection 2016 Mar-Apr. PMID 27104030
- [Background] N. G. Vailianou, A. Evangelopoulos, A. Kolia and C. Kazazis. Hypoglycemic and hipolipidemic effects of cinnamon. Current Topics in Nutraceutical Research. 2014;12(4):127-34
- [Background] Braissant O, Foufelle F, Scotto C, Dauca M, Wahli W. Differential expression of peroxisome proliferator-activated receptors (PPARs): tissue distribution of PPAR-alpha, -beta, and -gamma in the adult rat. Endocrinology. 1996 Jan;137(1):354-66. doi: 10.1210/endo.137.1.8536636.
- [Background] Sheng X, Zhang Y, Gong Z, Huang C, Zang YQ. Improved Insulin Resistance and Lipid Metabolism by Cinnamon Extract through Activation of Peroxisome Proliferator-Activated Receptors. PPAR Res. 2008;2008:581348. doi: 10.1155/2008/581348. Epub 2008 Dec 11. PMID 19096709
- [Background] Rao PV, Gan SH. Cinnamon: a multifaceted medicinal plant. Evid Based Complement Alternat Med. 2014;2014:642942. doi: 10.1155/2014/642942. Epub 2014 Apr 10. PMID 24817901
- [Background] Cao H, Polansky MM, Anderson RA. Cinnamon extract and polyphenols affect the expression of tristetraprolin, insulin receptor, and glucose transporter 4 in mouse 3T3-L1 adipocytes. Arch Biochem Biophys. 2007 Mar 15;459(2):214-22. doi: 10.1016/j.abb.2006.12.034. Epub 2007 Jan 25. PMID 17316549
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804
- [Background] Blevins SM, Leyva MJ, Brown J, Wright J, Scofield RH, Aston CE. Effect of cinnamon on glucose and lipid levels in non insulin-dependent type 2 diabetes. Diabetes Care. 2007 Sep;30(9):2236-7. doi: 10.2337/dc07-0098. Epub 2007 Jun 11. No abstract available. PMID 17563345
- [Background] Anderson RA, Zhan Z, Luo R, Guo X, Guo Q, Zhou J, Kong J, Davis PA, Stoecker BJ. Cinnamon extract lowers glucose, insulin and cholesterol in people with elevated serum glucose. J Tradit Complement Med. 2015 Apr 18;6(4):332-336. doi: 10.1016/j.jtcme.2015.03.005. eCollection 2016 Oct. PMID 27774415
- [Background] Lu T, Sheng H, Wu J, Cheng Y, Zhu J, Chen Y. Cinnamon extract improves fasting blood glucose and glycosylated hemoglobin level in Chinese patients with type 2 diabetes. Nutr Res. 2012 Jun;32(6):408-12. doi: 10.1016/j.nutres.2012.05.003. Epub 2012 Jun 14. PMID 22749176
- [Background] Hlebowicz J, Hlebowicz A, Lindstedt S, Bjorgell O, Hoglund P, Holst JJ, Darwiche G, Almer LO. Effects of 1 and 3 g cinnamon on gastric emptying, satiety, and postprandial blood glucose, insulin, glucose-dependent insulinotropic polypeptide, glucagon-like peptide 1, and ghrelin concentrations in healthy subjects. Am J Clin Nutr. 2009 Mar;89(3):815-21. doi: 10.3945/ajcn.2008.26807. Epub 2009 Jan 21. PMID 19158209
- [Background] R. A. Anderson. Cinnamon and Glucose Homeostasis. Nutrition Today. 2014;49(Supplement):S10-S1.
- [Background] E. E.-D. Gaber. Antidiabetic and hypolipidemic effects of Ceylon cinnamon (Cinnamomum verum) in alloxan-diabetic rats. Journal of Medicinal Plants Research 6(9): 1685-91, 2012.
- [Background] Allen RW, Schwartzman E, Baker WL, Coleman CI, Phung OJ. Cinnamon use in type 2 diabetes: an updated systematic review and meta-analysis. Ann Fam Med. 2013 Sep-Oct;11(5):452-9. doi: 10.1370/afm.1517. PMID 24019277
- [Background] A. S. Alanazi, M. U. Khan. Cinnamon use in type 2 diabetes an updated meta analysis. World Journal of Pharmacy and Pharmaceutical Sciences 4(05):1838-52, 2015.
- [Background] Costello RB, Dwyer JT, Saldanha L, Bailey RL, Merkel J, Wambogo E. Do Cinnamon Supplements Have a Role in Glycemic Control in Type 2 Diabetes? A Narrative Review. J Acad Nutr Diet. 2016 Nov;116(11):1794-1802. doi: 10.1016/j.jand.2016.07.015. Epub 2016 Sep 8. PMID 27618575
- [Background] Leach MJ, Kumar S. Cinnamon for diabetes mellitus. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007170. doi: 10.1002/14651858.CD007170.pub2. PMID 22972104
- [Background] Baker WL, Gutierrez-Williams G, White CM, Kluger J, Coleman CI. Effect of cinnamon on glucose control and lipid parameters. Diabetes Care. 2008 Jan;31(1):41-3. doi: 10.2337/dc07-1711. Epub 2007 Oct 1. PMID 17909085
- [Background] M. L. Casas Oñate and D. Montoya Martínez. ¿Son fiables los medidores de glucemia capilar?. Avances en Diabetología 28(5):110-3, 2012.
- [Background] I. Yépez, R. García and T. Toledo. Complicaciones agudas: Crisis hiperglucémica. Revista Venezolana de Endocrinología y Metabolismo 10:75-83, 2012.
- [Background] Pariente Rodrigo E, Deib-Morgan K, Garcia de Diego O, Garcia-Velasco P, Sgaramella GA, Garcia Gonzalez I. [Accuracy and reliability between glucose meters: A study under normal clinical practice conditions]. Semergen. 2017 Jan-Feb;43(1):20-27. doi: 10.1016/j.semerg.2016.01.011. Epub 2016 Mar 8. Spanish. PMID 26968861
- [Background] Dijkstra R, Braspenning J, Grol R. Empowering patients: how to implement a diabetes passport in hospital care. Patient Educ Couns. 2002 Jun;47(2):173-7. doi: 10.1016/s0738-3991(01)00196-3. PMID 12191541
- [Background] Azizi A, Aboutorabi R, Mazloum-Khorasani Z, Hoseini B, Tara M. Diabetic Personal Health Record: A Systematic Review Article. Iran J Public Health. 2016 Nov;45(11):1388-1398. PMID 28032056
- [Background] R. D. Cervantes-Villagrana and J. M. Presno-Bernal. Fisiopatología de la diabetes y los mecanismos de muerte de las células β pancreáticas. Revista de Endocrinología y Nutrición 21(3):98-106, 2013.
- [Result] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S55-S64. doi: 10.2337/dc18-S006. PMID 29222377
- [Result] Talaei B, Amouzegar A, Sahranavard S, Hedayati M, Mirmiran P, Azizi F. Effects of Cinnamon Consumption on Glycemic Indicators, Advanced Glycation End Products, and Antioxidant Status in Type 2 Diabetic Patients. Nutrients. 2017 Sep 8;9(9):991. doi: 10.3390/nu9090991. PMID 28885566
- [Result] Sami W, Ansari T, Butt NS, Hamid MRA. Effect of diet on type 2 diabetes mellitus: A review. Int J Health Sci (Qassim). 2017 Apr-Jun;11(2):65-71. PMID 28539866
- [Result] Davies MJ, Heller S, Skinner TC, Campbell MJ, Carey ME, Cradock S, Dallosso HM, Daly H, Doherty Y, Eaton S, Fox C, Oliver L, Rantell K, Rayman G, Khunti K; Diabetes Education and Self Management for Ongoing and Newly Diagnosed Collaborative. Effectiveness of the diabetes education and self management for ongoing and newly diagnosed (DESMOND) programme for people with newly diagnosed type 2 diabetes: cluster randomised controlled trial. BMJ. 2008 Mar 1;336(7642):491-5. doi: 10.1136/bmj.39474.922025.BE. Epub 2008 Feb 14. PMID 18276664
- [Result] Zare R, Nadjarzadeh A, Zarshenas MM, Shams M, Heydari M. Efficacy of cinnamon in patients with type II diabetes mellitus: A randomized controlled clinical trial. Clin Nutr. 2019 Apr;38(2):549-556. doi: 10.1016/j.clnu.2018.03.003. Epub 2018 Mar 11. PMID 29605574
- [Result] Azimi P, Ghiasvand R, Feizi A, Hosseinzadeh J, Bahreynian M, Hariri M, Khosravi-Boroujeni H. Effect of cinnamon, cardamom, saffron and ginger consumption on blood pressure and a marker of endothelial function in patients with type 2 diabetes mellitus: A randomized controlled clinical trial. Blood Press. 2016 Jun;25(3):133-40. doi: 10.3109/08037051.2015.1111020. Epub 2016 Jan 12. PMID 26758574
- [Result] Mahmoodnia L, Aghadavod E, Beigrezaei S, Rafieian-Kopaei M. An update on diabetic kidney disease, oxidative stress and antioxidant agents. J Renal Inj Prev. 2017 Jan 20;6(2):153-157. doi: 10.15171/jrip.2017.30. eCollection 2017. PMID 28497094
- [Result] Wei N, Zheng H, Nathan DM. Empirically establishing blood glucose targets to achieve HbA1c goals. Diabetes Care. 2014 Apr;37(4):1048-51. doi: 10.2337/dc13-2173. Epub 2014 Feb 10. PMID 24513588
- [Result] Klonoff DC. ADAG study group data links A1C levels with empirically measured blood glucose values - new treatment guidelines will now be needed. J Diabetes Sci Technol. 2014 May;8(3):439-43. doi: 10.1177/1932296814529638. Epub 2014 Apr 30. No abstract available. PMID 24876603
- [Result] Feller S, Boeing H, Pischon T. Body mass index, waist circumference, and the risk of type 2 diabetes mellitus: implications for routine clinical practice. Dtsch Arztebl Int. 2010 Jul;107(26):470-6. doi: 10.3238/arztebl.2010.0470. Epub 2010 Jul 2. PMID 20644701
- [Result] Funnell MM, Brown TL, Childs BP, Haas LB, Hosey GM, Jensen B, Maryniuk M, Peyrot M, Piette JD, Reader D, Siminerio LM, Weinger K, Weiss MA. National standards for diabetes self-management education. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S89-96. doi: 10.2337/dc10-S089. No abstract available. PMID 20042780
- See also: FDA - Substances Generally Recognized as Safe, Cinnamon bark, Ceylon. — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?fr=182.20.77
- See also: FDA - Compliance Policy Guides (CPGs), CPG Sec. 525.750 Spices - Definitions, 10. Cinnamon — https://www.fda.gov/iceci/compliancemanuals/compliancepolicyguidancemanual/ucm074468.htm
- See also: Diabetes Atlas, International Federation of Diabetes — http://www.diabetesatlas.org/
- See also: World Health Organization. World report on diabetes 2016 — http://apps.who.int/iris/bitstream/10665/254649/1/9789243565255-spa.pdf